CLINICAL TRIAL: NCT02907736
Title: Impact of Neutrophil Extracellular Traps on Tissue Plasminogen Activator Induced Thrombolysis in Acute Ischemic Stroke Patients
Acronym: THROMBONETS
Status: Withdrawn | Type: Observational
Why Stopped: replaced by a new study
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JDS_2015_45
Record Dates: First submitted 2016-09-06; First posted 2016-09-20 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Acute Ischemic stroke (AIS) remains a leading cause of adult disability, cognitive impairment and mortality worldwide despite the development of revascularization therapies (intravenous Tissue Plasminogen Activator (t-PA) and endovascular therapy). Thrombosis resistance after IV t-PA therapy is frequent especially in case of AIS with proximal occlusion. In recent years, neutrophil extracellular traps (NETs) have been identified as major triggers and structural factors of various forms of thrombosis. NETs are extracellular webs primarily composed of DNA from neutrophils. A recent study shows that the NETs burden in coronary thrombi is positively correlated with the infarct size and negatively correlated with electrocardiogram (ST-segment) resolution. This later study revealed that in vitro addition of DNase I accelerated the t-PA-induced thrombolysis of coronary thrombi. NETs could, in consequence, be promising targets for improved thrombolysis in AIS.

The aim of this study is to assess the impact of NETs composition of thrombi retrieved during endovascular therapy in AIS patients on IV t-PA induced thrombolysis, clinical outcome and AIS etiologies.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* AIS secondary to a large vessel occlusion
* admitted for endovascular therapy.

Exclusion Criteria:

* Pregnant or breast feeding patient patient under legal protection
* Patient opposition to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute stroke, admitted for endovascular therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
thrombus origin | baseline
  according to the etiology of the stroke (TOAST classification)
red cells counts | baseline
  quantitative assessment of the relative fractions of the main constituents after Hematoxylin and Eosin staining :
white cells counts | baseline
  quantitative assessment of the relative fractions of the main constituents after Hematoxylin and Eosin staining
platlet counts | baseline
  quantitative assessment of the relative fractions of the main constituents after Hematoxylin and Eosin staining

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Désilles, MD, Principal Investigator — Fondation OPH A. de Rothschild; Mikael Mazighi, MD, PhD, Study Chair — Fondation OPH A. de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France

REFERENCES:
- [Derived] Ducroux C, Di Meglio L, Loyau S, Delbosc S, Boisseau W, Deschildre C, Ben Maacha M, Blanc R, Redjem H, Ciccio G, Smajda S, Fahed R, Michel JB, Piotin M, Salomon L, Mazighi M, Ho-Tin-Noe B, Desilles JP. Thrombus Neutrophil Extracellular Traps Content Impair tPA-Induced Thrombolysis in Acute Ischemic Stroke. Stroke. 2018 Mar;49(3):754-757. doi: 10.1161/STROKEAHA.117.019896. Epub 2018 Feb 8. PMID 29438080